CLINICAL TRIAL: NCT03991286
Title: The Effect of Astaxanthin on Oxidative Stress Indices in Serum, and Induction of Signaling Pathways in Granulosa Cells in Patients With Polycystic Ovary Syndrome
Brief Title: The Effect of Astaxanthin on Oxidative Stress Indices in Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 98-01-30-41687
Record Dates: First submitted 2019-05-22; First posted 2019-06-19 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2020-02

CONDITIONS: PCOS
Keywords: PCOS; Astaxanthin; ROS
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Drug: Placebo
  Ovulatory Agent:
  Clomiphene Citrate
  Interventions: Other: placebo
- experimental (Experimental): Drug: Astaxanthin 8mg
  Drug: Ovulatory Agent Clomiphene Citrate
  Interventions: Dietary Supplement: Astaxanthin 8 mg

INTERVENTIONS:
Dietary Supplement: Astaxanthin 8 mg — experimental
  Other Names: Algalife, Icelandic Astaxanthin
  Arms: experimental
Other: placebo — Matching placebo pill
  Arms: Placebo

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy affecting women of reproductive age It is hypothesized that ∼20 fold increase in reactive oxygen species (ROS) generation in Follicular fluid (FF) and granulosa cells of PCOS women plays an adverse role in affecting the IVF success rate. Astaxanthin (3,3'-dihydroxy-β,β'-carotene-4,4'-dione) is a nonprovitamin A carotenoid classified as a xanthophyll and is found in high amounts in the red pigment of crustacean shells (e.g., crabs, shrimp), salmon, trout, and asteroides. It has been demonstrated that astaxanthin displays a wide variety of biological activities, including anti-oxidative, anticancer, and anti-inflammatory effects.

investigators aim to investigate the effect on Astaxanthin administrating on reducing of ROS in FF and induction of antioxidant response elements in PCOS women.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed PCOS cases according to the National Institute of Health criteria (NIH consensus criteria) and Rotterdam criteria

Exclusion Criteria:

* Menopause, pregnant or lactating females
* individuals with diabetes
* those with hepatic,renal, thyroid or cardiovascular disorders
* patients with elevated levels of prolactin
* those who were taking antioxidant supplements within the last 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Serum and follicular fluid oxidative stress biomarkers levels | 8 months
  This parameter will measure using Enzyme-Linked. Immunosorbent Assays (ELISAs)

SECONDARY OUTCOMES:
Number of oocytes retrieved | Day1(from the day of oocyte retrieval to fertilization confirmation)
  using polarized light microscopy
Number of mature(MII) oocyte | Day1(from the day of oocyte retrieval to fertilization confirmation)
  using polarized light microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Fardin Amidi, professor, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Shariati Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gharaei R, Alyasin A, Mahdavinezhad F, Samadian E, Ashrafnezhad Z, Amidi F. Randomized controlled trial of astaxanthin impacts on antioxidant status and assisted reproductive technology outcomes in women with polycystic ovarian syndrome. J Assist Reprod Genet. 2022 Apr;39(4):995-1008. doi: 10.1007/s10815-022-02432-0. Epub 2022 Mar 3. PMID 35237893